CLINICAL TRIAL: NCT02216123
Title: A Randomized, Double-Blind, Double Dummy, Comparative, Multicenter Study to Assess the Incidence of Hemolysis, Safety, and Efficacy of Tafenoquine (SB-252263, WR238605) Versus Primaquine in the Treatment of Subjects With Plasmodium Vivax Malaria
Brief Title: Study to Assess the Incidence of Hemolysis, Safety, and Efficacy of Tafenoquine (SB-252263, WR238605) Versus Primaquine in Subjects With Plasmodium Vivax Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116564
Record Dates: First submitted 2014-06-19; First posted 2014-08-13 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-02

CONDITIONS: Malaria, Vivax
Keywords: Tafenoquine; Plasmodium vivax; Hemolysis; Primaquine; Chloroquine; Glucose-6-phosphate dehydrogenase (G6PD); Relapse
MeSH Terms: conditions — Malaria, Vivax; Hemolysis; Recurrence | interventions — tafenoquine; Chloroquine; Primaquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tafenoquine+ Chloroquine (Experimental): All subjects will receive one of two formulations of CQ from Days 1 to 3 (600 mg [2×CQ 300 mg] on Day 1, 600 mg on Day 2 and 300 mg on Day 3, each once daily [OD] orally; OR, 620 mg [4×CQ 155 mg] on Day 1, 620 mg on Day 2 and 310 mg on Day 3, each once daily [OD] orally). Tafenoquine 300mg (2×TQ 150 mg) will be given as a single oral dose on Day 1 or Day 2. Primaquine matching placebo will be given OD orally beginning on Day 1 or Day 2 and continue for 14 days total dosing. All subjects will be followed-up till 180 days.
  Interventions: Drug: Tafenoquine; Drug: Chloroquine; Drug: Primaquine Placebo
- Primaquine+ Chloroquine (Experimental): All subjects will receive one of two formulations of CQ from Days 1 to 3 (600 mg [2×CQ 300 mg] on Day 1, 600 mg on Day 2 and 300 mg on Day 3, each once daily [OD] orally; OR, 620 mg [4×CQ 155 mg] on Day 1, 620 mg on Day 2 and 310 mg on Day 3, each once daily [OD] orally). Primaquine 15mg will be given OD orally beginning on Day 1 or Day 2 and continue for 14 total dosing. Tafenoquine matching placebo will be given as a single oral dose on Day 1 or Day 2. All subjects will be followed-up till 180 days.
  Interventions: Drug: Tafenoquine Placebo; Drug: Chloroquine; Drug: Primaquine

INTERVENTIONS:
Drug: Tafenoquine — Tafenoquine will be supplied as a dark pink, capsule-shaped, film-coated tablet that is plain on both sides. Each tablet will contain 150mg TQ.
  Arms: Tafenoquine+ Chloroquine
Drug: Tafenoquine Placebo — Placebo TQ tablets will be supplied as a dark pink, capsule-shaped, film-coated tablet that is plain on both sides, with common excipients of appropriate quality.
  Arms: Primaquine+ Chloroquine
Drug: Chloroquine — One of two formulations of commercially available generic chloroquine may be utilized in this study:
  1. tablets containing 500 mg chloroquine phosphate (equivalent to 300 mg chloroquine free base); or,
  2. tablets containing 250 mg chloroquine phosphate (equivalent to 155 mg chloroquine free base).
Drug: Primaquine — Commercially available primaquine containing primaquine phosphate united states pharmacopeia (USP), 26.3 mg (equivalent to primaquine base 15 mg) will be utilized in this study. Primaquine, a pink film-coated tablet imprinted W on one side and P97 on the other side. The PQ tablets for this study have been over-encapsulated in a Swedish orange size B supro capsule.
  Arms: Primaquine+ Chloroquine
Drug: Primaquine Placebo — Placebo to match PQ will be supplied as Swedish orange size B supro capsules with common excipients of appropriate quality.
  Arms: Tafenoquine+ Chloroquine

SUMMARY:
This is a prospective, double-blind, double-dummy, multicenter, comparative study. A total of 300 subjects will be randomized to treatment on Day 1, of which a minimum of 50 female subjects must be enrolled that display moderate glucose-6-phosphate dehydrogenase (G6PD) deficiency (>=40% - <70% of the site median G6PD value). Subjects must have a blood smear that is positive for P. vivax at entry. Subjects will be randomized 2:1 to receive tafenoquine (TQ)/chloroquine(CQ) or the active comparator primaquine (PQ)/CQ. All subjects will receive CQ on Days 1 to 3, followed by TQ or PQ and matching placebo beginning on Day 1 or 2. Tafenoquine, or matching placebo, will be given as a single, 300mg dose. Subjects will receive PQ (15mg once daily) or matching placebo for 14 days. The duration of the study is 180 days, including screening and randomization to treatment (Day 1), three in-hospital days (Days 1-3), four out-patient visits while on treatment with study medication (Days 5, 8, 11 and 15) and seven follow-up visits (Days 22, 29, 60, 90, 120, 150 and 180).

The primary safety data collected in this study will help to understand the hemolysis risk to both G6PD-normal and G6PD-deficient subjects. The efficacy data produced from this study will support the results for sister study TAF112582, the pivotal phase III efficacy and safety study of the TQ program.

ELIGIBILITY:
Inclusion Criteria:

* A female is eligible to enter and participate in the study if she is non-pregnant, nonlactating and if she is of: a. Non-childbearing potential defined as: post-menopausal (12 months of spontaneous amenorrhea or <6 months of spontaneous amenorrhea with serum follicle-stimulating hormone >40 milli-International units per milliliter [mIU/mL]), or pre-menopausal and has had a hysterectomy or a bilateral oophorectomy (removal of the ovaries) or a bilateral tubal ligation, negative pregnancy test or, b. Child-bearing potential, has a negative pregnancy test at screening, and agrees to comply with one of the following during the treatment stage of the study and for a period of 90 days after stopping study medication: Use of oral contraceptive, either combined or progestogen alone used in conjunction with double barrier method as defined below. Use of an intrauterine device with a documented failure rate of <1% per year; Use of depo provera injection; Double barrier method consisting of spermicide with either condom or diaphragm; Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female. Complete abstinence from intercourse for 2 weeks prior to administration of study medication, throughout the study and for a period of 90 days after stopping study medication.
* The subject has a glucose 6-phosphate dehydrogenase (G6PD) value (measured by a quantitative spectrophotometric phenotype assay) as follows: Female subjects must have an enzyme level >= 40 percent of the site median value for G6PD normal males. Male subjects must have an enzyme level >= 70 percent of the site median value for G6PD normal males.
* The subject has a screening hemoglobin (Hb) value as follows: Any subject with a G6PD value >=70 percent of the site median value must have a screening Hb value >=7 g/dL; Female subjects with a G6PD value is >=40 - <70 percent of the site median value must have a screening Hb value >=8 g/dL.
* The subject has a QT duration corrected for heart rate by Fridericia's Formula (QTcF) <450 milisecond (msec). Reading based on an average of triplicate Electrocardiograms (ECGs) obtained over a brief recording period by machine or manual over-read.
* The subject has a positive malarial smear for P. vivax .
* The subject has a parasite density of >100 and <100,000 per microliter (μL).
* Male or female subject aged 16 years or older (18 years or older in Ethiopia) at the time of signing the informed consent.
* The subject agrees to G6PD genotyping.
* The subject is willing and able to comply with the study protocol.
* The subject or parent/legal guardian, as applicable, has given written informed, dated consent; and the subject has given written assent, if applicable, to participate in the study.

Exclusion Criteria:

* The subject has a mixed malaria infection (identified by a malarial smear or rapid diagnostic test).
* The subject has severe P. vivax malaria as defined by World Health Organization (WHO) criteria.
* The subject has a history of allergy to chloroquine, mefloquine, tafenoquine, primaquine, or to any other 4- or 8-aminoquinoline.
* The subject has a liver alanine aminotransferase (ALT) >2 x upper limit of normal (ULN).
* The subject has severe vomiting (no food or inability to take food during the previous 8 hours).
* The subject has a clinically significant concurrent illness (e.g., pneumonia, septicemia), pre-existing condition (e.g., renal disease, malignancy), condition that may affect absorption of study medication (e.g., vomiting, severe diarrhea), or clinical signs and symptoms of severe cardiovascular disease (e.g., uncontrolled congestive heart failure, severe coronary artery disease).
* The subject has a history of porphyria, psoriasis, or epilepsy.
* The subject has a history of significant ocular disease (e.g. surgery to the globe, glaucoma, diabetic retinopathy) or has evidence of corneal or retinal abnormalities identified in the clinical screening ophthalmologic examination.
* The subject has taken anti-malarials (e.g., artemisinin-based combination therapies, mefloquine, primaquine, or any other 4- or 8-aminoquinoline) within 30 days prior to study entry.
* The subject has taken or will likely require during the study the use of medications from the following classes: Histamine-2 blockers and antacids; Drugs with hemolytic potential; Drugs known to prolong the QTcF interval; The biguanides phenformin and buformin (but excluding metformin); Drugs that are substrates of the renal transporters OCT2, MATE1 AND MATE-2K and have a narrow therapeutic index (for example, the anti-arrhythmic agents dofetilide, procainamide and pilsicainide)
* The subject has received treatment with any investigational drug within 30 days of study entry, or within 5 half-lives, whichever is longer.
* The subject has a recent history of illicit drug abuse or heavy alcohol intake, such that full participation in the study could be compromised.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- GSK Investigational Site, Manaus, Amazonas, Brazil
- Colombia (2):
  - GSK Investigational Site, Cali
  - GSK Investigational Site, Montería
- Ethiopia (2):
  - GSK Investigational Site, Gonder
  - GSK Investigational Site, Jimma
- GSK Investigational Site, Iquitos, Loreto, Peru
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Mae Sot
  - GSK Investigational Site, Tak
- GSK Investigational Site, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Llanos-Cuentas A, Lacerda MVG, Hien TT, Velez ID, Namaik-Larp C, Chu CS, Villegas MF, Val F, Monteiro WM, Brito MAM, Costa MRF, Chuquiyauri R, Casapia M, Nguyen CH, Aruachan S, Papwijitsil R, Nosten FH, Bancone G, Angus B, Duparc S, Craig G, Rousell VM, Jones SW, Hardaker E, Clover DD, Kendall L, Mohamed K, Koh GCKW, Wilches VM, Breton JJ, Green JA. Tafenoquine versus Primaquine to Prevent Relapse of Plasmodium vivax Malaria. N Engl J Med. 2019 Jan 17;380(3):229-241. doi: 10.1056/NEJMoa1802537. PMID 30650326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized, double-blind, double-dummy, comparative, multicenter study to assess the incidence of hemolysis, safety and efficacy of Tafenoquine (TQ) versus Primaquine (PQ) in treatment of participants with Plasmodium vivax (P. vivax) malaria.
Pre-assignment Details: A total of 369 participants were screened of which 118 failed screening and 251 participants were randomized to receive either TQ+chloroquine (CQ) or PQ+CQ in a ratio of 2:1.
Groups:
- TQ+CQ: Participants were administered CQ 600 milligram (mg) once daily on Days 1 and 2 and CQ 300 mg on Day 3. A single dose of TQ 300 mg was administered orally on Day 1 or Day 2. PQ placebo capsules were administered orally once daily for 14 days starting on the same day as TQ administration.
- PQ+CQ: Participants were administered CQ 600 mg tablet once daily on Days 1 and 2 and CQ 300 mg on Day 3. Participants received a single TQ placebo tablet orally on Day 1 or Day 2. PQ 15 mg was administered orally once daily for 14 days starting on the same day as TQ placebo administration.
Period: Overall Study
Arm/Group | TQ+CQ | PQ+CQ
Started | 166 | 85
Completed | 160 | 83
Not Completed | 6 | 2
Not completed — Lost to Follow-up | 4 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TQ+CQ | PQ+CQ | Total
Number analyzed (Participants) | 166 | 85 | 251
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.5 (14.28) | 37.7 (14.69) | 37.6 (14.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 32 | 84
  Male | 114 | 53 | 167
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  American (Amer) Indian (Ind) or Alaska Native (N) | 87 | 43 | 130
  Asian-East Asian Heritage | 6 | 3 | 9
  Asian-South East Asian Heritage | 35 | 20 | 55
  Black or African Amer | 2 | 0 | 2
  African Amer/African Heritage/Amer Ind or Alaska N | 36 | 19 | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Relevant Hemolysis.
Description: Clinically relevant hemolysis is defined as a decrease in hemoglobin of >=30% or >3 grams per deciliter (g/dL) from Baseline; or, an overall drop in hemoglobin below 6.0 g/dL at any visit after the first dose of study medication. The percentage of participants with clinically relevant hemolysis has been summarized. Safety Population comprised of all randomized participants who received at least one dose of blinded study medication.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Percentage of participants | 2.41 [0.941 to 6.031] | 1.18 [0.208 to 6.367]
Statistical Analysis 1: Comparison: TQ+CQ vs PQ+CQ; Test type: Other; Mean Difference (Final Values) = 1.23, 95% CI 2-sided [-4.161 to 4.982] — Confidence interval for the treatment difference was based on the Newcombe method. Percent treatment difference (TQ+CQ-PQ+CQ) has been presented

2. Primary Outcome: Percentage of Female Participants With Moderate Glucose-6 Phosphate Dehydrogenase (G6PD) Deficiency Experiencing Clinically Relevant Hemolysis.
Description: Clinically relevant hemolysis is defined as a decrease in hemoglobin of >=30% or >3 g/dL from Baseline; or, an overall drop in hemoglobin below 6.0 g/dL at any visit after the first dose of study medication. Despite additional efforts, no females with moderate G6PD-deficiency were enrolled that experienced clinically-significant hemolysis during the study; hence, the end point could not be estimated.
Time Frame: Up to Day 180
Population: Safety Population
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Rate of Relapse-free Efficacy at Six Months Post Dose
Description: A participant was considered to have demonstrated relapse-free efficacy at 6 months if: a) Participant had non-zero P. vivax asexual parasite count at Baseline. b) Participant showed initial clearance of P. vivax parasitemia defined as two negative asexual P. vivax parasite counts, with at least 6 hours between the counts, and no positive counts in the interval. c) Participant had no positive asexual P. vivax parasite count at any assessment prior to or on Study Day 201 following initial parasite clearance. d) Participant did not take a concomitant medication with anti-malarial activity at any point between Study Day 1 and their last parasite assessment. e) Participant is parasite-free at 6 months. The rate of relapse-free efficacy was estimated by Kaplan-Meier methodology. The percentage of participants who were relapse-free at 6 months post dose has been presented along with 95% confidence interval.
Time Frame: 6 months post dose
Population: Microbiologic-Intent-To-Treat (mITT) Population comprised of all randomized participants who received at least one dose of blinded study medication and had microscopically-confimed P. vivax parasitemia at Baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Percentage of participants | 72.7 [64.8 to 79.2] | 75.1 [64.2 to 83.2]
Statistical Analysis 1: Comparison: TQ+CQ vs PQ+CQ; Test type: Other; Hazard Ratio (HR) = 0.984, 95% CI [0.577 to 1.678] — Hazards ratio was estimated from Cox Proportional Hazards Model with treatment and region as covariates. A hazard ratio <1 indicates a lower chance of relapse with TQ+CQ compared to PQ+CQ

4. Secondary Outcome: Rate of Relapse-free Efficacy at Four Months Post Dose
Description: A participant was considered to have demonstrated recurrence-free efficacy at 4 months if: a) Participant had non-zero P. vivax asexual parasite count at Baseline. b) Participant showed initial clearance of P. vivax parasitemia. c) Participant had no positive asexual P. vivax parasite count at any assessment prior to or on Study Day 130 following initial parasite clearance. d) Participant did not take a concomitant medication with anti-malarial activity at any point between Study Day 1 and their last parasite assessment after Study Day 109 (up to and including Study Day 130). e) Participant is parasite-free at 4 months. The rate of relapse-free efficacy was estimated by Kaplan-Meier methodology. The percentage of participants who were relapse-free at 4 months post dose has been presented along with 95% confidence interval.
Time Frame: 4 months post dose
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Percentage of participants | 82.3 [74.9 to 87.7] | 79.7 [68.9 to 87.1]
Statistical Analysis 1: Comparison: TQ+CQ vs PQ+CQ; Test type: Other; Hazard Ratio (HR) = 0.815, 95% CI 2-sided [0.442 to 1.503] — Hazard ratio was estimated from Cox Proportional Hazards Model with treatment and region as covariates. A hazard ratio<1 indicates a lower chance of relapse with TQ+CQ compared to PQ+CQ

5. Secondary Outcome: Time to Relapse of P. Vivax Malaria
Description: Relapse is defined by a positive blood smear with or without vivax symptoms. Relapse is described as any recurrence of malaria that occurred after Day 32 of the study. The time to relapse was analyzed by the Kaplan-Meier method. The median number of days to relapse along with 95% confidence interval has been presented for each treatment group.
Time Frame: Up to Day 180
Population: mITT Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Days | NA [NA to NA] — The median estimate for the time to relapse is the time taken (in days) for 50% of participants to relapse. As less than 50% of participants in both treatment arms relapsed during the study, the median times to relapse could not be calculated. | NA [NA to NA] — The median estimate for the time to relapse is the time taken (in days) for 50% of participants to relapse. As less than 50% of participants in both treatment arms relapsed during the study, the median times to relapse could not be calculated.

6. Secondary Outcome: Time to Parasite Clearance
Description: Parasite clearance time is defined as time needed to clear asexual parasite from the blood that is, parasite numbers falling below the limit of detection in the thick blood smear and remaining undetectable after 6 to 12 hours later. The time to achieve parasite clearance was analyzed by Kaplan-Meier methodology. The median parasite clearance time along with 95% confidence interval has been presented for each treatment group.
Time Frame: Up to Day 180
Population: mITT Population
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Hours | 41 [38 to 45] | 44 [41 to 49]

7. Secondary Outcome: Time to Fever Clearance
Description: Fever clearance time is defined as the time from first dose of treatment to the time when body temperature falls to normal within Study Days 1-4 and remains normal for at least 48 hours up to the Day 8 visit. Fever clearance was considered to have been achieved once an initial temperature of more than 37.4 degree Celsius is reduced to a value less than or equal to 37.4 degree Celsius, in the absence of value more than 37.4 degree Celsius in the following 48 hours up to the Day 8 visit. The time taken to achieve fever clearance was analyzed by Kaplan-Meier method.
Time Frame: Up to Day 9
Population: mITT Population
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Hours | 10 [7 to 19] | 13 [8 to 22]

8. Secondary Outcome: Time to Gametocyte Clearance
Description: Gametocyte clearance time is defined as time from first dose until the first slide that was gametocyte negative and remained so at the next slide reading. The time taken to achieve gametocyte clearance was analyzed by Kaplan-Meier method.
Time Frame: Up to Day 180
Population: mITT Population
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Hours | 38 [37 to 43] | 41 [37 to 48]

9. Secondary Outcome: Number of Participants With Recrudescence
Description: Recrudescence is defined as any P. vivax parasitemia occurring on or before Day 32 (that is, blood stage treatment failure). A participant was considered to have had a recrudescence if both of the following were true: a) Participant had a positive P. vivax asexual parasite count at Baseline and demonstrated clearance (that is, did not have two negative asexual P. vivax parasite counts, with at least 6 hours between the counts, and no positive counts in the interval). b) Participant had a positive genetically homologous asexual P. vivax parasite count, after their zero count in Days 1 to 5, but on or before Study Day 32. The number of participants with recrudescence before Study Day 33 has been presented.
Time Frame: Up to Day 32
Population: mITT Population
Measure: Number; unit: Participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Genetically Homologous and Genetically Heterologous P. Vivax Infections
Description: Two drops of peripheral blood were collected onto pre-printed filter paper for subsequent deoxyribonucleic acid (DNA) extraction and polymerase chain reaction (PCR) analysis of Plasmodium species on all participants at screening (Day 1; pre-dose) and; if necessary, at the time of the first recrudescence/relapse or re-infection. PCR of the P. vivax genes, was used to distinguish between genetically homologous and genetically heterologous infection. The number of participants with genetically homologous and genetically heterologous P. vivax infections has been summarized for each treatment group. Only those participants with an infection occuring on or after Study Day 33 were analyzed.
Time Frame: Up to Day 180
Population: mITT Population. Only those participants who had a recurrence of infection were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 42 | 20
Participants
  Heterologous P. vivax | 8 | 9
  Homologous P. vivax | 29 | 10
  Unknown genetic classification | 5 | 1

11. Secondary Outcome: Number of Participants With Clinical Chemistry Laboratory Data Outside the Reference Range
Description: Plasma or serum samples were anlalyzed to evaluate clinical chemistry parameters such as alanine aminotransferase (ALT), alkaline phosphatase (ALP), aspartate aminotransferase (AST), bilirubin, creatine kinase, creatinine, glomerular filtration rate (GFR), indirect bilirubin and urea. The number of participants with clinical chemistry laboratory values outside the extended normal range (F3) has been presented. The upper and lower limits for F3 range were defined by multiplying the normal range limits by different factors. High and low indicated that the participants had values flagged as high and low respectively for the particular parameter any time on-treatment. Safety Population consisted of all randomized participants who received at least one dose of blinded study medication.
Time Frame: Up to Day 120
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Participants
  ALT, High | 8 | 0
  ALP, High | 0 | 1
  AST, High | 6 | 3
  Bilirubin, High | 28 | 18
  Creatine kinase, High | 3 | 4
  Creatinine, High | 0 | 0
  GFR, Low | 0 | 0
  Indirect bilirubin, High | 36 | 21
  Urea, High | 40 | 19

12. Secondary Outcome: Number of Participants With Hematology Laboratory Data Outside the Reference Range
Description: Blood samples were collected for the evaluation of hematology parameters including eosinophils, leukocytes, lymphocytes, neutrophils, platelets, reticulocytes and methemoglobin. The number of participants with hematology laboratory data outside the extended normal range (F3) has been presented. The upper and lower limits for F3 range were defined by multiplying the normal range limits by different factors. High and low indicated that the participants had values flagged as high and low respectively for the particular parameter any time on-treatment. Participants having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters were counted in both the High and Low categories.
Time Frame: Up to Day 120
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Participants
  Blood eosinophils, High | 32 | 15
  Blood leukocytes, Low | 0 | 0
  Blood lymphocytes, Low | 8 | 1
  Blood lymphocytes, High | 11 | 4
  Blood neutrophils, Low | 5 | 3
  Blood platelets, Low | 13 | 8
  Blood reticulocytes, High | 80 | 39
  Methemoglobin, High | 2 | 3

13. Secondary Outcome: Number of Participants With Abnormal Urinalysis Dipstick Results
Description: Mid-stream urine was collected and analyzed for bilirubin, glucose, ketones, leukocyte esterase (LE), nitrites, occult blood, proteins and urobilinogen by dipstick method. The number of participants with abnormal urinalysis results (Trace, +, ++, +++, ++++) has been presented. Only those participants with data available at the specified data points were analyzed.
Time Frame: Up to Day 120
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Participants
  Bilirubin, Day 1, Trace: number analyzed (Participants) | 166 | 84
  Bilirubin, Day 1, Trace | 1 | 1
  Bilirubin, Day 1, +: number analyzed (Participants) | 166 | 84
  Bilirubin, Day 1, + | 9 | 2
  Bilirubin, Day1, ++: number analyzed (Participants) | 166 | 84
  Bilirubin, Day1, ++ | 3 | 0
  Bilirubin, Day 3, +: number analyzed (Participants) | 165 | 85
  Bilirubin, Day 3, + | 8 | 3
  Bilirubin, Day 3, ++: number analyzed (Participants) | 165 | 85
  Bilirubin, Day 3, ++ | 2 | 0
  Bilirubin, Day 5, Trace | 1 | 0
  Bilirubin, Day 5, + | 4 | 0
  Bilirubin, Day 8, +: number analyzed (Participants) | 164 | 84
  Bilirubin, Day 8, + | 0 | 2
  Bilirubin, Day 11, Trace: number analyzed (Participants) | 163 | 84
  Bilirubin, Day 11, Trace | 1 | 1
  Bilirubin, Day 22, Trace: number analyzed (Participants) | 164 | 84
  Bilirubin, Day 22, Trace | 0 | 1
  Bilirubin, Day 22, +: number analyzed (Participants) | 164 | 84
  Bilirubin, Day 22, + | 1 | 0
  Bilirubin, Day 60, Trace: number analyzed (Participants) | 160 | 83
  Bilirubin, Day 60, Trace | 0 | 1
  Bilirubin, Day 60, +: number analyzed (Participants) | 160 | 83
  Bilirubin, Day 60, + | 2 | 1
  Bilirubin, Day 90, +: number analyzed (Participants) | 160 | 82
  Bilirubin, Day 90, + | 0 | 1
  Bilirubin, Day 120, +: number analyzed (Participants) | 160 | 81
  Bilirubin, Day 120, + | 3 | 2
  Glucose, Day 1, +: number analyzed (Participants) | 166 | 84
  Glucose, Day 1, + | 2 | 1
  Glucose, Day 1, ++: number analyzed (Participants) | 166 | 84
  Glucose, Day 1, ++ | 0 | 1
  Glucose, Day1, +++: number analyzed (Participants) | 166 | 84
  Glucose, Day1, +++ | 2 | 3
  Glucose, Day1, ++++: number analyzed (Participants) | 166 | 84
  Glucose, Day1, ++++ | 0 | 1
  Glucose, Day 3, +: number analyzed (Participants) | 165 | 85
  Glucose, Day 3, + | 0 | 1
  Glucose, Day 3, ++: number analyzed (Participants) | 165 | 85
  Glucose, Day 3, ++ | 1 | 1
  Glucose, Day 3, +++: number analyzed (Participants) | 165 | 85
  Glucose, Day 3, +++ | 0 | 2
  Glucose, Day 3, ++++: number analyzed (Participants) | 165 | 85
  Glucose, Day 3, ++++ | 0 | 1
  Glucose, Day 5, ++ | 0 | 1
  Glucose, Day 5, +++ | 0 | 3
  Glucose, Day 8, +: number analyzed (Participants) | 164 | 84
  Glucose, Day 8, + | 1 | 1
  Glucose, Day 8, ++: number analyzed (Participants) | 164 | 84
  Glucose, Day 8, ++ | 0 | 1
  Glucose, Day 8,+++: number analyzed (Participants) | 164 | 84
  Glucose, Day 8,+++ | 0 | 1
  Glucose, Day 11, Trace: number analyzed (Participants) | 163 | 84
  Glucose, Day 11, Trace | 0 | 1
  Glucose, Day 11, +: number analyzed (Participants) | 163 | 84
  Glucose, Day 11, + | 0 | 2
  Glucose, Day 11, ++: number analyzed (Participants) | 163 | 84
  Glucose, Day 11, ++ | 3 | 0
  Glucose, Day 11, +++: number analyzed (Participants) | 163 | 84
  Glucose, Day 11, +++ | 1 | 1
  Glucose, Day 15, ++: number analyzed (Participants) | 165 | 84
  Glucose, Day 15, ++ | 0 | 1
  Glucose, Day 15, +++: number analyzed (Participants) | 165 | 84
  Glucose, Day 15, +++ | 1 | 0
  Glucose, Day 15, ++++: number analyzed (Participants) | 165 | 84
  Glucose, Day 15, ++++ | 0 | 1
  Glucose, Day 22, +: number analyzed (Participants) | 164 | 84
  Glucose, Day 22, + | 1 | 2
  Glucose, Day 22, +++: number analyzed (Participants) | 164 | 84
  Glucose, Day 22, +++ | 0 | 1
  Glucose, Day 29, Trace: number analyzed (Participants) | 162 | 84
  Glucose, Day 29, Trace | 1 | 0
  Glucose, Day 29, ++: number analyzed (Participants) | 162 | 84
  Glucose, Day 29, ++ | 1 | 2
  Glucose, Day 60, +: number analyzed (Participants) | 160 | 83
  Glucose, Day 60, + | 0 | 4
  Glucose, Day 60, ++: number analyzed (Participants) | 160 | 83
  Glucose, Day 60, ++ | 1 | 1
  Glucose, Day 90, +: number analyzed (Participants) | 160 | 82
  Glucose, Day 90, + | 0 | 1
  Glucose, Day 90, ++: number analyzed (Participants) | 160 | 82
  Glucose, Day 90, ++ | 0 | 1
  Glucose, Day 90, +++: number analyzed (Participants) | 160 | 82
  Glucose, Day 90, +++ | 1 | 1
  Glucose, Day 120, Trace: number analyzed (Participants) | 160 | 81
  Glucose, Day 120, Trace | 1 | 0
  Glucose, Day 120, +: number analyzed (Participants) | 160 | 81
  Glucose, Day 120, + | 1 | 1
  Glucose, Day 120, ++: number analyzed (Participants) | 160 | 81
  Glucose, Day 120, ++ | 0 | 2
  Glucose, Day 120, +++: number analyzed (Participants) | 160 | 81
  Glucose, Day 120, +++ | 0 | 2
  Glucose, Day 120, ++++: number analyzed (Participants) | 160 | 81
  Glucose, Day 120, ++++ | 1 | 0
  Ketones, Day 1, Trace: number analyzed (Participants) | 166 | 84
  Ketones, Day 1, Trace | 3 | 0
  Ketones, Day 1, +: number analyzed (Participants) | 166 | 84
  Ketones, Day 1, + | 4 | 2
  Ketones, Day1, ++: number analyzed (Participants) | 166 | 84
  Ketones, Day1, ++ | 4 | 3
  Ketones, Day1, +++: number analyzed (Participants) | 166 | 84
  Ketones, Day1, +++ | 2 | 1
  Ketones, Day 3, Trace: number analyzed (Participants) | 165 | 85
  Ketones, Day 3, Trace | 0 | 1
  Ketones, Day 3, +: number analyzed (Participants) | 165 | 85
  Ketones, Day 3, + | 5 | 3
  Ketones, Day 3, ++: number analyzed (Participants) | 165 | 85
  Ketones, Day 3, ++ | 3 | 2
  Ketones, Day 3, +++: number analyzed (Participants) | 165 | 85
  Ketones, Day 3, +++ | 3 | 0
  Ketones, Day 5, + | 1 | 0
  Ketones, Day 8, +: number analyzed (Participants) | 164 | 84
  Ketones, Day 8, + | 1 | 1
  Ketones, Day 11, Trace: number analyzed (Participants) | 163 | 84
  Ketones, Day 11, Trace | 1 | 0
  Ketones, Day 22, Trace: number analyzed (Participants) | 164 | 84
  Ketones, Day 22, Trace | 1 | 1
  Ketones, Day 22, +: number analyzed (Participants) | 164 | 84
  Ketones, Day 22, + | 1 | 0
  Ketones, Day 90, Trace: number analyzed (Participants) | 160 | 82
  Ketones, Day 90, Trace | 2 | 0
  Ketones, Day 90, +: number analyzed (Participants) | 160 | 82
  Ketones, Day 90, + | 0 | 1
  Ketones, Day 90, ++: number analyzed (Participants) | 160 | 82
  Ketones, Day 90, ++ | 1 | 0
  Ketones, Day 120, Trace: number analyzed (Participants) | 160 | 81
  Ketones, Day 120, Trace | 1 | 0
  Ketones, Day 120, +: number analyzed (Participants) | 160 | 81
  Ketones, Day 120, + | 1 | 0
  Ketones, Day 120, ++: number analyzed (Participants) | 160 | 81
  Ketones, Day 120, ++ | 1 | 0
  LE, Day 1, Trace: number analyzed (Participants) | 166 | 84
  LE, Day 1, Trace | 3 | 1
  LE, Day 1, +: number analyzed (Participants) | 166 | 84
  LE, Day 1, + | 19 | 9
  LE, Day1, ++: number analyzed (Participants) | 166 | 84
  LE, Day1, ++ | 5 | 2
  LE, Day1, +++: number analyzed (Participants) | 166 | 84
  LE, Day1, +++ | 1 | 2
  LE, Day 3, Trace: number analyzed (Participants) | 165 | 85
  LE, Day 3, Trace | 4 | 0
  LE, Day 3, +: number analyzed (Participants) | 165 | 85
  LE, Day 3, + | 13 | 5
  LE, Day 3, ++: number analyzed (Participants) | 165 | 85
  LE, Day 3, ++ | 2 | 1
  LE, Day 3, +++: number analyzed (Participants) | 165 | 85
  LE, Day 3, +++ | 1 | 0
  LE, Day 5, Trace: number analyzed (Participants) | 165 | 85
  LE, Day 5, Trace | 3 | 1
  LE, Day 5, +: number analyzed (Participants) | 165 | 85
  LE, Day 5, + | 11 | 4
  LE, Day 5, ++: number analyzed (Participants) | 165 | 85
  LE, Day 5, ++ | 3 | 2
  LE, Day 5, +++: number analyzed (Participants) | 165 | 85
  LE, Day 5, +++ | 3 | 2
  LE, Day 8, Trace: number analyzed (Participants) | 164 | 84
  LE, Day 8, Trace | 7 | 3
  LE, Day 8, +: number analyzed (Participants) | 164 | 84
  LE, Day 8, + | 10 | 4
  LE, Day 8, ++: number analyzed (Participants) | 164 | 84
  LE, Day 8, ++ | 6 | 1
  LE, Day 8, +++: number analyzed (Participants) | 164 | 84
  LE, Day 8, +++ | 2 | 2
  LE, Day 11, Trace: number analyzed (Participants) | 163 | 84
  LE, Day 11, Trace | 6 | 2
  LE, Day 11, +: number analyzed (Participants) | 163 | 84
  LE, Day 11, + | 11 | 3
  LE, Day 11, ++: number analyzed (Participants) | 163 | 84
  LE, Day 11, ++ | 3 | 3
  LE, Day 11, +++: number analyzed (Participants) | 163 | 84
  LE, Day 11, +++ | 3 | 1
  LE, Day 15, Trace: number analyzed (Participants) | 165 | 84
  LE, Day 15, Trace | 8 | 2
  LE, Day 15, +: number analyzed (Participants) | 165 | 84
  LE, Day 15, + | 4 | 8
  LE, Day 15, ++: number analyzed (Participants) | 165 | 84
  LE, Day 15, ++ | 4 | 3
  LE, Day 15, +++: number analyzed (Participants) | 165 | 84
  LE, Day 15, +++ | 2 | 1
  LE, Day 22, Trace: number analyzed (Participants) | 164 | 84
  LE, Day 22, Trace | 4 | 2
  LE, Day 22, +: number analyzed (Participants) | 164 | 84
  LE, Day 22, + | 13 | 4
  LE, Day 22, ++: number analyzed (Participants) | 164 | 84
  LE, Day 22, ++ | 3 | 0
  LE, Day 22, +++: number analyzed (Participants) | 164 | 84
  LE, Day 22, +++ | 1 | 1
  LE, Day 29, Trace: number analyzed (Participants) | 162 | 84
  LE, Day 29, Trace | 5 | 0
  LE, Day 29, +: number analyzed (Participants) | 162 | 84
  LE, Day 29, + | 11 | 6
  LE, Day 29, ++: number analyzed (Participants) | 162 | 84
  LE, Day 29, ++ | 1 | 4
  LE, Day 29, +++: number analyzed (Participants) | 162 | 84
  LE, Day 29, +++ | 4 | 0
  LE, Day 60, Trace: number analyzed (Participants) | 160 | 83
  LE, Day 60, Trace | 8 | 3
  LE, Day 60, +: number analyzed (Participants) | 160 | 83
  LE, Day 60, + | 8 | 4
  LE, Day 60, ++: number analyzed (Participants) | 160 | 83
  LE, Day 60, ++ | 5 | 2
  LE, Day 60, +++: number analyzed (Participants) | 160 | 83
  LE, Day 60, +++ | 2 | 1
  LE, Day 90, Trace: number analyzed (Participants) | 159 | 82
  LE, Day 90, Trace | 6 | 1
  LE, Day 90, +: number analyzed (Participants) | 159 | 82
  LE, Day 90, + | 13 | 7
  LE, Day 90, ++: number analyzed (Participants) | 159 | 82
  LE, Day 90, ++ | 2 | 2
  LE, Day 90, +++: number analyzed (Participants) | 159 | 82
  LE, Day 90, +++ | 0 | 1
  LE, Day 120, Trace: number analyzed (Participants) | 160 | 81
  LE, Day 120, Trace | 5 | 1
  LE, Day 120, +: number analyzed (Participants) | 160 | 81
  LE, Day 120, + | 12 | 3
  LE, Day 120, ++: number analyzed (Participants) | 160 | 81
  LE, Day 120, ++ | 5 | 2
  LE, Day 120, +++: number analyzed (Participants) | 160 | 81
  LE, Day 120, +++ | 0 | 1
  Nitrite, Day 1, Trace: number analyzed (Participants) | 166 | 84
  Nitrite, Day 1, Trace | 1 | 0
  Nitrite, Day 1, +: number analyzed (Participants) | 166 | 84
  Nitrite, Day 1, + | 4 | 0
  Nitrite, Day 3, +: number analyzed (Participants) | 165 | 85
  Nitrite, Day 3, + | 1 | 0
  Nitrite, Day 5, + | 1 | 0
  Nitrite, Day 5, +++ | 1 | 0
  Nitrite, Day 8, +++: number analyzed (Participants) | 164 | 84
  Nitrite, Day 8, +++ | 1 | 0
  Nitrite, Day 11, +: number analyzed (Participants) | 163 | 84
  Nitrite, Day 11, + | 1 | 1
  Nitrite, Day 15, +: number analyzed (Participants) | 165 | 84
  Nitrite, Day 15, + | 2 | 0
  Nitrite, Day 22, Trace: number analyzed (Participants) | 164 | 84
  Nitrite, Day 22, Trace | 1 | 0
  Nitrite, Day 29, +: number analyzed (Participants) | 162 | 84
  Nitrite, Day 29, + | 2 | 0
  Nitrite, Day 60, +: number analyzed (Participants) | 160 | 83
  Nitrite, Day 60, + | 3 | 0
  Nitrite, Day 90, Trace: number analyzed (Participants) | 160 | 82
  Nitrite, Day 90, Trace | 0 | 1
  Nitrite, Day 90, +: number analyzed (Participants) | 160 | 82
  Nitrite, Day 90, + | 2 | 1
  Nitrite, Day 120, +: number analyzed (Participants) | 160 | 81
  Nitrite, Day 120, + | 2 | 1
  Nitrite, Day 120, ++: number analyzed (Participants) | 160 | 81
  Nitrite, Day 120, ++ | 1 | 0
  Occult blood, Day 1, Trace | 2 | 4
  Occult blood, Day 1, + | 18 | 7
  Occult blood, Day 1, ++ | 9 | 4
  Occult blood, Day1, +++ | 12 | 2
  Occult blood, Day1, ++++ | 6 | 1
  Occult blood, Day 3, Trace: number analyzed (Participants) | 165 | 85
  Occult blood, Day 3, Trace | 4 | 3
  Occult blood, Day 3, +: number analyzed (Participants) | 165 | 85
  Occult blood, Day 3, + | 14 | 6
  Occult blood, Day 3, ++: number analyzed (Participants) | 165 | 85
  Occult blood, Day 3, ++ | 9 | 3
  Occult blood, Day 3, +++: number analyzed (Participants) | 165 | 85
  Occult blood, Day 3, +++ | 5 | 3
  Occult blood, Day 3, ++++: number analyzed (Participants) | 165 | 85
  Occult blood, Day 3, ++++ | 3 | 1
  Occult blood, Day 5, Trace | 4 | 1
  Occult blood, Day 5, + | 7 | 3
  Occult blood, Day 5, ++ | 6 | 3
  Occult blood, Day 5, +++ | 4 | 2
  Occult blood, Day 5, ++++ | 3 | 2
  Occult blood, Day 8, Trace: number analyzed (Participants) | 164 | 84
  Occult blood, Day 8, Trace | 4 | 4
  Occult blood, Day 8, +: number analyzed (Participants) | 164 | 84
  Occult blood, Day 8, + | 12 | 4
  Occult blood, Day 8, ++: number analyzed (Participants) | 164 | 84
  Occult blood, Day 8, ++ | 3 | 0
  Occult blood, Day 8,+++: number analyzed (Participants) | 164 | 84
  Occult blood, Day 8,+++ | 3 | 2
  Occult blood, Day 11, Trace: number analyzed (Participants) | 163 | 84
  Occult blood, Day 11, Trace | 2 | 1
  Occult blood, Day 11, +: number analyzed (Participants) | 163 | 84
  Occult blood, Day 11, + | 8 | 3
  Occult blood, Day 11, ++: number analyzed (Participants) | 163 | 84
  Occult blood, Day 11, ++ | 3 | 2
  Occult blood, Day 11, +++: number analyzed (Participants) | 163 | 84
  Occult blood, Day 11, +++ | 3 | 0
  Occult blood, Day 11, ++++: number analyzed (Participants) | 163 | 84
  Occult blood, Day 11, ++++ | 1 | 1
  Occult blood, Day 15, Trace: number analyzed (Participants) | 165 | 84
  Occult blood, Day 15, Trace | 2 | 1
  Occult blood, Day 15, +: number analyzed (Participants) | 165 | 84
  Occult blood, Day 15, + | 11 | 2
  Occult blood, Day 15, ++: number analyzed (Participants) | 165 | 84
  Occult blood, Day 15, ++ | 3 | 2
  Occult blood, Day 15, +++: number analyzed (Participants) | 165 | 84
  Occult blood, Day 15, +++ | 2 | 1
  Occult blood, Day 15, ++++: number analyzed (Participants) | 165 | 84
  Occult blood, Day 15, ++++ | 0 | 1
  Occult blood, Day 22, Trace: number analyzed (Participants) | 164 | 84
  Occult blood, Day 22, Trace | 4 | 1
  Occult blood, Day 22, +: number analyzed (Participants) | 164 | 84
  Occult blood, Day 22, + | 11 | 5
  Occult blood, Day 22, ++: number analyzed (Participants) | 164 | 84
  Occult blood, Day 22, ++ | 4 | 1
  Occult blood, Day 22, +++: number analyzed (Participants) | 164 | 84
  Occult blood, Day 22, +++ | 2 | 1
  Occult blood, Day 22, ++++: number analyzed (Participants) | 164 | 84
  Occult blood, Day 22, ++++ | 1 | 1
  Occult blood, Day 29, Trace: number analyzed (Participants) | 162 | 84
  Occult blood, Day 29, Trace | 5 | 2
  Occult blood, Day 29, +: number analyzed (Participants) | 162 | 84
  Occult blood, Day 29, + | 17 | 5
  Occult blood, Day 29, ++: number analyzed (Participants) | 162 | 84
  Occult blood, Day 29, ++ | 3 | 1
  Occult blood, Day 29, +++: number analyzed (Participants) | 162 | 84
  Occult blood, Day 29, +++ | 3 | 4
  Occult blood, Day 29, ++++: number analyzed (Participants) | 162 | 84
  Occult blood, Day 29, ++++ | 1 | 0
  Occult blood, Day 60, Trace: number analyzed (Participants) | 160 | 83
  Occult blood, Day 60, Trace | 5 | 0
  Occult blood, Day 60, +: number analyzed (Participants) | 160 | 83
  Occult blood, Day 60, + | 15 | 7
  Occult blood, Day 60, ++: number analyzed (Participants) | 160 | 83
  Occult blood, Day 60, ++ | 2 | 3
  Occult blood, Day 60, +++: number analyzed (Participants) | 160 | 83
  Occult blood, Day 60, +++ | 3 | 0
  Occult blood, Day 60, ++++: number analyzed (Participants) | 160 | 83
  Occult blood, Day 60, ++++ | 1 | 0
  Occult blood, Day 90, Trace: number analyzed (Participants) | 160 | 82
  Occult blood, Day 90, Trace | 4 | 1
  Occult blood, Day 90, +: number analyzed (Participants) | 160 | 82
  Occult blood, Day 90, + | 13 | 7
  Occult blood, Day 90, ++: number analyzed (Participants) | 160 | 82
  Occult blood, Day 90, ++ | 7 | 2
  Occult blood, Day 90, +++: number analyzed (Participants) | 160 | 82
  Occult blood, Day 90, +++ | 4 | 3
  Occult blood, Day 90, ++++: number analyzed (Participants) | 160 | 82
  Occult blood, Day 90, ++++ | 2 | 2
  Occult blood, Day 120, Trace: number analyzed (Participants) | 160 | 81
  Occult blood, Day 120, Trace | 2 | 2
  Occult blood, Day 120, +: number analyzed (Participants) | 160 | 81
  Occult blood, Day 120, + | 13 | 5
  Occult blood, Day 120, ++: number analyzed (Participants) | 160 | 81
  Occult blood, Day 120, ++ | 3 | 3
  Occult blood, Day 120, +++: number analyzed (Participants) | 160 | 81
  Occult blood, Day 120, +++ | 6 | 0
  Occult blood, Day 120, ++++: number analyzed (Participants) | 160 | 81
  Occult blood, Day 120, ++++ | 0 | 2
  Protein, Day 1, Trace | 15 | 8
  Protein, Day 1, + | 19 | 8
  Protein, Day1, ++ | 4 | 1
  Protein, Day 3, Trace: number analyzed (Participants) | 165 | 85
  Protein, Day 3, Trace | 8 | 6
  Protein, Day 3, +: number analyzed (Participants) | 165 | 85
  Protein, Day 3, + | 21 | 13
  Protein, Day 3, ++: number analyzed (Participants) | 165 | 85
  Protein, Day 3, ++ | 3 | 1
  Protein, Day 5, Trace | 5 | 5
  Protein, Day 5, + | 4 | 1
  Protein, Day 5, ++ | 2 | 1
  Protein, Day 8, Trace: number analyzed (Participants) | 164 | 84
  Protein, Day 8, Trace | 6 | 4
  Protein, Day 8, +: number analyzed (Participants) | 164 | 84
  Protein, Day 8, + | 6 | 2
  Protein, Day 8,++: number analyzed (Participants) | 164 | 84
  Protein, Day 8,++ | 1 | 0
  Protein, Day 11, Trace: number analyzed (Participants) | 163 | 84
  Protein, Day 11, Trace | 1 | 3
  Protein, Day 11, +: number analyzed (Participants) | 163 | 84
  Protein, Day 11, + | 4 | 1
  Protein, Day 11, ++: number analyzed (Participants) | 163 | 84
  Protein, Day 11, ++ | 1 | 0
  Protein, Day 15, +: number analyzed (Participants) | 165 | 84
  Protein, Day 15, + | 2 | 0
  Protein, Day 15, ++: number analyzed (Participants) | 165 | 84
  Protein, Day 15, ++ | 1 | 0
  Protein, Day 22, Trace: number analyzed (Participants) | 164 | 84
  Protein, Day 22, Trace | 2 | 1
  Protein, Day 22, +: number analyzed (Participants) | 164 | 84
  Protein, Day 22, + | 2 | 1
  Protein, Day 22, ++: number analyzed (Participants) | 164 | 84
  Protein, Day 22, ++ | 1 | 0
  Protein, Day 29, Trace: number analyzed (Participants) | 162 | 84
  Protein, Day 29, Trace | 3 | 1
  Protein, Day 29, +: number analyzed (Participants) | 162 | 84
  Protein, Day 29, + | 4 | 0
  Protein, Day 29, ++: number analyzed (Participants) | 162 | 84
  Protein, Day 29, ++ | 1 | 0
  Protein, Day 60, Trace: number analyzed (Participants) | 160 | 83
  Protein, Day 60, Trace | 3 | 1
  Protein, Day 60, +: number analyzed (Participants) | 160 | 83
  Protein, Day 60, + | 3 | 2
  Protein, Day 60, ++: number analyzed (Participants) | 160 | 83
  Protein, Day 60, ++ | 1 | 0
  Protein, Day 90, Trace: number analyzed (Participants) | 160 | 82
  Protein, Day 90, Trace | 4 | 1
  Protein Day 90, +: number analyzed (Participants) | 160 | 82
  Protein Day 90, + | 3 | 0
  Protein, Day 120, Trace: number analyzed (Participants) | 160 | 81
  Protein, Day 120, Trace | 2 | 1
  Protein, Day 120, +: number analyzed (Participants) | 160 | 81
  Protein, Day 120, + | 6 | 0
  Protein, Day 120, ++: number analyzed (Participants) | 160 | 81
  Protein, Day 120, ++ | 1 | 0
  Urobilinogen, Day 1, Trace: number analyzed (Participants) | 166 | 84
  Urobilinogen, Day 1, Trace | 8 | 0
  Urobilinogen, Day 1, +: number analyzed (Participants) | 166 | 84
  Urobilinogen, Day 1, + | 23 | 5
  Urobilinogen, Day1, ++: number analyzed (Participants) | 166 | 84
  Urobilinogen, Day1, ++ | 10 | 4
  Urobilinogen, Day1, +++: number analyzed (Participants) | 166 | 84
  Urobilinogen, Day1, +++ | 3 | 1
  Urobilinogen, Day 3, Trace: number analyzed (Participants) | 165 | 85
  Urobilinogen, Day 3, Trace | 6 | 2
  Urobilinogen, Day 3, +: number analyzed (Participants) | 165 | 85
  Urobilinogen, Day 3, + | 14 | 11
  Urobilinogen, Day 3, ++: number analyzed (Participants) | 165 | 85
  Urobilinogen, Day 3, ++ | 8 | 4
  Urobilinogen Day 3, +++: number analyzed (Participants) | 165 | 85
  Urobilinogen Day 3, +++ | 0 | 3
  Urobilinogen, Day 3, ++++: number analyzed (Participants) | 165 | 85
  Urobilinogen, Day 3, ++++ | 0 | 1
  Urobilinogen, Day 5, Trace | 3 | 1
  Urobilinogen, Day 5, + | 3 | 2
  Urobilinogen, Day 8, Trace: number analyzed (Participants) | 164 | 84
  Urobilinogen, Day 8, Trace | 2 | 2
  Urobilinogen, Day 8, +: number analyzed (Participants) | 164 | 84
  Urobilinogen, Day 8, + | 0 | 2
  Urobilinogen, Day 8, ++: number analyzed (Participants) | 164 | 84
  Urobilinogen, Day 8, ++ | 0 | 1
  Urobilinogen, Day 8,+++: number analyzed (Participants) | 164 | 84
  Urobilinogen, Day 8,+++ | 0 | 1
  Urobilinogen, Day 11, Trace: number analyzed (Participants) | 163 | 84
  Urobilinogen, Day 11, Trace | 1 | 1
  Urobilinogen, Day 11, +: number analyzed (Participants) | 163 | 84
  Urobilinogen, Day 11, + | 2 | 0
  Urobilinogen, Day 11, ++: number analyzed (Participants) | 163 | 84
  Urobilinogen, Day 11, ++ | 0 | 1
  Urobilinogen, Day 15, Trace: number analyzed (Participants) | 164 | 84
  Urobilinogen, Day 15, Trace | 3 | 1
  Urobilinogen, Day 15, +: number analyzed (Participants) | 164 | 84
  Urobilinogen, Day 15, + | 1 | 0
  Urobilinogen, Day 15, ++: number analyzed (Participants) | 164 | 84
  Urobilinogen, Day 15, ++ | 1 | 0
  Urobilinogen, Day 22, Trace: number analyzed (Participants) | 164 | 84
  Urobilinogen, Day 22, Trace | 3 | 0
  Urobilinogen, Day 29, Trace: number analyzed (Participants) | 162 | 84
  Urobilinogen, Day 29, Trace | 4 | 1
  Urobilinogen, Day 29, +: number analyzed (Participants) | 162 | 84
  Urobilinogen, Day 29, + | 2 | 1
  Urobilinogen, Day 60, Trace: number analyzed (Participants) | 160 | 83
  Urobilinogen, Day 60, Trace | 3 | 1
  Urobilinogen, Day 60, +: number analyzed (Participants) | 160 | 83
  Urobilinogen, Day 60, + | 1 | 0
  Urobilinogen, Day 90, Trace: number analyzed (Participants) | 160 | 82
  Urobilinogen, Day 90, Trace | 4 | 1
  Urobilinogen, Day 90, +: number analyzed (Participants) | 160 | 82
  Urobilinogen, Day 90, + | 3 | 0
  Urobilinogen, Day 120, Trace: number analyzed (Participants) | 160 | 81
  Urobilinogen, Day 120, Trace | 2 | 0
  Urobilinogen, Day 120, +: number analyzed (Participants) | 160 | 81
  Urobilinogen, Day 120, + | 2 | 0
  Urobilinogen, Day 120, ++: number analyzed (Participants) | 160 | 81
  Urobilinogen, Day 120, ++ | 0 | 1

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant under clinical investigation, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/ birth defect, other situations such as important medical events and events of possible drug induced liver injury with hyperbilirubinemia. TEAEs are defined as AEs with an onset date and time on or after that of the start of first dose of study medication (including CQ). Number of participants with TEAEs and serious TEAEs have been presented.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Participants
  TEAEs | 119 | 64
  Serious TEAEs | 6 | 1

15. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Findings
Description: 12 lead ECG was performed with the participant in a semi-supine position having rested in this position for at least 10 minutes. ECG assessments were performed in triplicate at screening followed by single ECGs 12 hours after the first dose of study medication and at Day 29. The number of participants with abnormal-clinically significant ECG findings have been presented. The 12 Hour Post Randomized Treatment (11.5-12.5 Hours) timepoint included all readings taken between 11.5 and 12.5 hours post randomized treatment. The 12 Hour Post Randomized Treatment (8-72 Hours) timepoint is a sensitivity analysis of the 12 Hour post randomized treatment timepoint, including all readings taken between 8 and 72 hours post randomized treatment. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Day 29
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Participants
  11.5 to 12.5 hours Day 1, Assessment 1; n=143, 75: number analyzed (Participants) | 143 | 75
  11.5 to 12.5 hours Day 1, Assessment 1; n=143, 75 | 0 | 0
  11.5 to 12.5 hours Day 1 Assessment 2; n=6, 6: number analyzed (Participants) | 6 | 6
  11.5 to 12.5 hours Day 1 Assessment 2; n=6, 6 | 0 | 0
  11.5 to 12.5 hours Day 1 Assessment 3; n=5, 5: number analyzed (Participants) | 5 | 5
  11.5 to 12.5 hours Day 1 Assessment 3; n=5, 5 | 0 | 0
  8 to 72 hours Day 1 Assessment 1; n=166, 85 | 0 | 0
  8 to 72 hours Day 1 Assessment 2; n=6, 6: number analyzed (Participants) | 6 | 6
  8 to 72 hours Day 1 Assessment 2; n=6, 6 | 0 | 0
  8 to 72 hours Day 1 Assessment 3; n=5, 5: number analyzed (Participants) | 5 | 5
  8 to 72 hours Day 1 Assessment 3; n=5, 5 | 0 | 0
  Day 29; n=161, 84: number analyzed (Participants) | 161 | 84
  Day 29; n=161, 84 | 0 | 0

16. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) and Mean Arterial Pressure (MAP)
Description: Vital signs were measured twice a day on Days 1 through 3, at least 4 hours apart, and immediately prior to pharmacokinetic (PK) measurements. MAP was calculated as the sum of SBP and two times DBP divided by 3. The mean and standard deviation of SBP, DBP and MAP has been presented. The values presented does not include Day 3 assessments for participant number 570. Baseline value is defined as the latest pre-treatment assessment where treatment is their first dose of study medication (CQ/PQ/TQ/Placebo). Change from Baseline is the value at post dose minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Day 180
Population: Safety Population
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
millimeter of mercury (mmHg)
  SBP, Day 1 assessment 4; n=161, 84: number analyzed (Participants) | 161 | 84
  SBP, Day 1 assessment 4; n=161, 84 | 1.2 (10.98) | -0.9 (10.73)
  SBP, Day 2 assessment 1; n=166, 85 | 0.4 (11.78) | -2.3 (10.91)
  SBP, Day 2 assessment 4; n=166, 85 | -0.8 (12.21) | -2.7 (12.46)
  SBP, Day 3 assessment 1; n=166, 83: number analyzed (Participants) | 166 | 83
  SBP, Day 3 assessment 1; n=166, 83 | -0.6 (13.38) | -2.1 (11.69)
  SBP, Day 3 assessment 4; n=166, 82: number analyzed (Participants) | 166 | 82
  SBP, Day 3 assessment 4; n=166, 82 | -2.7 (12.45) | -2.2 (12.66)
  SBP, Day 8; n=164, 84: number analyzed (Participants) | 164 | 84
  SBP, Day 8; n=164, 84 | 2.2 (12.00) | 0.8 (12.47)
  SBP, Day 11; n=163, 84: number analyzed (Participants) | 163 | 84
  SBP, Day 11; n=163, 84 | 1.3 (12.35) | 1.2 (14.69)
  SBP, Day15; n=165, 84: number analyzed (Participants) | 165 | 84
  SBP, Day15; n=165, 84 | 3.2 (13.81) | 2.5 (12.64)
  SBP, Day 22; n=164, 84: number analyzed (Participants) | 164 | 84
  SBP, Day 22; n=164, 84 | 3.3 (13.21) | 2.9 (12.55)
  SBP, Day 29; n=163, 84: number analyzed (Participants) | 163 | 84
  SBP, Day 29; n=163, 84 | 2.6 (14.08) | 4.4 (14.29)
  SBP, Day 60; n=160, 83: number analyzed (Participants) | 160 | 83
  SBP, Day 60; n=160, 83 | 4.4 (14.10) | 4.3 (15.95)
  SBP, Day 90; n=160, 82: number analyzed (Participants) | 160 | 82
  SBP, Day 90; n=160, 82 | 3.8 (14.30) | 5.3 (14.91)
  SBP, Day 120; n=159, 81: number analyzed (Participants) | 159 | 81
  SBP, Day 120; n=159, 81 | 3.8 (14.05) | 3.1 (15.40)
  SBP, Day 150; n=161, 82: number analyzed (Participants) | 161 | 82
  SBP, Day 150; n=161, 82 | 4.4 (13.99) | 4.9 (12.83)
  SBP, Day180; n=160, 83: number analyzed (Participants) | 160 | 83
  SBP, Day180; n=160, 83 | 3.7 (14.21) | 5.7 (13.64)
  DBP, Day 1 assessment 4; n=161, 84: number analyzed (Participants) | 161 | 84
  DBP, Day 1 assessment 4; n=161, 84 | 1.1 (7.56) | -1.5 (8.07)
  DBP, Day 2 assessment 1; n=166, 85 | -0.1 (8.67) | -2.2 (8.42)
  DBP, Day 2 assessment 4; n=166, 85 | -0.8 (9.57) | -2.6 (8.99)
  DBP, Day 3 assessment 1; n=166, 83: number analyzed (Participants) | 166 | 83
  DBP, Day 3 assessment 1; n=166, 83 | -0.2 (10.91) | -1.3 (9.28)
  DBP, Day 3 assessment 4; n=166, 82: number analyzed (Participants) | 166 | 82
  DBP, Day 3 assessment 4; n=166, 82 | -1.9 (9.69) | -1.9 (9.79)
  DBP, Day 8; n=164, 84: number analyzed (Participants) | 164 | 84
  DBP, Day 8; n=164, 84 | 0.9 (8.93) | 1.1 (9.99)
  DBP, Day 11; n=163, 84: number analyzed (Participants) | 163 | 84
  DBP, Day 11; n=163, 84 | -0.0 (9.42) | -0.5 (9.39)
  DBP, Day15; n=165, 84: number analyzed (Participants) | 165 | 84
  DBP, Day15; n=165, 84 | 1.5 (10.91) | 0.4 (9.74)
  DBP, Day 22; n=164, 84: number analyzed (Participants) | 164 | 84
  DBP, Day 22; n=164, 84 | 1.2 (10.00) | 1.3 (9.25)
  DBP, Day 29; n=163, 84: number analyzed (Participants) | 163 | 84
  DBP, Day 29; n=163, 84 | 0.9 (10.58) | 1.5 (10.79)
  DBP, Day 60; n=160, 83: number analyzed (Participants) | 160 | 83
  DBP, Day 60; n=160, 83 | 3.1 (11.05) | 1.9 (10.34)
  DBP, Day 90; n=160, 82: number analyzed (Participants) | 160 | 82
  DBP, Day 90; n=160, 82 | 2.7 (11.60) | 3.5 (9.32)
  DBP, Day 120; n=159, 81: number analyzed (Participants) | 159 | 81
  DBP, Day 120; n=159, 81 | 3.3 (10.99) | 2.4 (10.83)
  DBP, Day 150; n=161, 82: number analyzed (Participants) | 161 | 82
  DBP, Day 150; n=161, 82 | 3.2 (11.15) | 4.1 (10.96)
  DBP, Day180; n=160, 83: number analyzed (Participants) | 160 | 83
  DBP, Day180; n=160, 83 | 2.9 (11.04) | 3.7 (10.71)
  MAP, Day 1 assessment 4; n=161, 84: number analyzed (Participants) | 161 | 84
  MAP, Day 1 assessment 4; n=161, 84 | 1.1 (7.45) | -1.3 (7.98)
  MAP, Day 2 assessment 1; n=166, 85 | 0.0 (8.68) | -2.2 (8.08)
  MAP, Day 2 assessment 4; n=166, 85 | -0.8 (9.48) | -2.6 (9.14)
  MAP, Day 3 assessment 1; n=166, 83: number analyzed (Participants) | 166 | 83
  MAP, Day 3 assessment 1; n=166, 83 | -0.3 (10.75) | -1.6 (8.98)
  MAP, Day 3 assessment 4; n=166, 82: number analyzed (Participants) | 166 | 82
  MAP, Day 3 assessment 4; n=166, 82 | -2.2 (9.76) | -2.0 (9.91)
  MAP, Day 8; n=164, 84: number analyzed (Participants) | 164 | 84
  MAP, Day 8; n=164, 84 | 1.3 (8.98) | 1.0 (9.76)
  MAP, Day 11; n=163, 84: number analyzed (Participants) | 163 | 84
  MAP, Day 11; n=163, 84 | 0.4 (9.33) | 0.1 (9.51)
  MAP, Day15; n=165, 84: number analyzed (Participants) | 165 | 84
  MAP, Day15; n=165, 84 | 2.0 (10.72) | 1.1 (9.58)
  MAP, Day 22; n=164, 84: number analyzed (Participants) | 164 | 84
  MAP, Day 22; n=164, 84 | 1.9 (9.94) | 1.8 (9.06)
  MAP, Day 29; n=163, 84: number analyzed (Participants) | 163 | 84
  MAP, Day 29; n=163, 84 | 1.5 (10.58) | 2.4 (10.80)
  MAP, Day 60; n=160, 83: number analyzed (Participants) | 160 | 83
  MAP, Day 60; n=160, 83 | 3.5 (11.07) | 2.7 (10.79)
  MAP, Day 90; n=160, 82: number analyzed (Participants) | 160 | 82
  MAP, Day 90; n=160, 82 | 3.1 (11.34) | 4.1 (9.76)
  MAP, Day 120; n=159, 81: number analyzed (Participants) | 159 | 81
  MAP, Day 120; n=159, 81 | 3.5 (10.66) | 2.6 (10.90)
  MAP, Day 150; n=161, 82: number analyzed (Participants) | 161 | 82
  MAP, Day 150; n=161, 82 | 3.6 (10.83) | 4.4 (10.44)
  MAP, Day180; n=160, 83: number analyzed (Participants) | 160 | 83
  MAP, Day180; n=160, 83 | 3.2 (10.91) | 4.4 (9.95)

17. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Vital signs were measured twice a day on Days 1 through 3, at least 4 hours apart, and immediately prior to PK measurements. The mean and standard deviation of pulse rate has been presented. The values presented does not include Day 3 assessments for participant number 570. Baseline value is defined as the latest pre-treatment assessment where treatment is their first dose of study medication (CQ/PQ/TQ/Placebo). Change from Baseline is the value at post dose minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Day 180
Population: Safety Population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
beats per minute
  Day 1 assessment 4; n=161, 84: number analyzed (Participants) | 161 | 84
  Day 1 assessment 4; n=161, 84 | -10.8 (15.24) | -9.3 (15.05)
  Day 2 assessment 1; n=166, 85 | -9.9 (17.06) | -9.9 (14.90)
  Day 2 assessment 4; n=166, 85 | -11.9 (15.78) | -11.8 (13.74)
  Day 3 assessment 1; n=166, 83: number analyzed (Participants) | 166 | 83
  Day 3 assessment 1; n=166, 83 | -15.1 (16.62) | -18.2 (16.09)
  Day 3 assessment 4; n=166, 82: number analyzed (Participants) | 166 | 82
  Day 3 assessment 4; n=166, 82 | -16.5 (17.16) | -17.5 (16.17)
  Day 8; n=164, 84: number analyzed (Participants) | 164 | 84
  Day 8; n=164, 84 | -12.7 (16.49) | -14.6 (17.91)
  Day 11; n=163, 84: number analyzed (Participants) | 163 | 84
  Day 11; n=163, 84 | -13.4 (17.83) | -15.5 (17.05)
  Day15; n=165, 84: number analyzed (Participants) | 165 | 84
  Day15; n=165, 84 | -13.5 (17.98) | -16.9 (17.77)
  Day 22; n=164, 84: number analyzed (Participants) | 164 | 84
  Day 22; n=164, 84 | -14.7 (17.72) | -16.8 (17.08)
  Day 29; n=163, 84: number analyzed (Participants) | 163 | 84
  Day 29; n=163, 84 | -16.9 (16.85) | -17.5 (16.27)
  Day 60; n=160, 83: number analyzed (Participants) | 160 | 83
  Day 60; n=160, 83 | -16.7 (17.44) | -18.5 (17.51)
  Day 90; n=160, 82: number analyzed (Participants) | 160 | 82
  Day 90; n=160, 82 | -16.3 (16.87) | -18.6 (17.27)
  Day 120; n=159, 81: number analyzed (Participants) | 159 | 81
  Day 120; n=159, 81 | -16.7 (17.82) | -19.1 (18.40)
  Day 150; n=161, 82: number analyzed (Participants) | 161 | 82
  Day 150; n=161, 82 | -16.8 (16.60) | -17.9 (18.32)
  Day180; n=160, 83: number analyzed (Participants) | 160 | 83
  Day180; n=160, 83 | -18.0 (18.51) | -18.3 (18.27)

18. Secondary Outcome: Change From Baseline in Temperature
Description: Vital signs were performed twice a day on Days 1 through 3, at least 4 hours apart, and immediately prior to PK measurements. The mean and standard deviation of pulse rate has been presented. The values presented does not include Day 3 assessments for participant number 570. Baseline value is defined as the latest pre-treatment assessment where treatment is their first dose of study medication (CQ/PQ/TQ/Placebo). Change from Baseline is the value at post dose minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Day 180
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Celsius
  Day 1 assessment 4; n=161, 84: number analyzed (Participants) | 161 | 84
  Day 1 assessment 4; n=161, 84 | -0.6 (1.05) | -0.5 (1.29)
  Day 2 assessment 1; n=166, 85 | -0.6 (1.20) | -0.6 (1.36)
  Day 2 assessment 4; n=166, 85 | -0.6 (1.08) | -0.6 (1.14)
  Day 3 assessment 1; n=166, 83: number analyzed (Participants) | 166 | 83
  Day 3 assessment 1; n=166, 83 | -1.0 (1.03) | -0.9 (1.10)
  Day 3 assessment 4; n=166, 82: number analyzed (Participants) | 166 | 82
  Day 3 assessment 4; n=166, 82 | -1.0 (1.02) | -1.0 (1.09)
  Day 8; n=164, 84: number analyzed (Participants) | 164 | 84
  Day 8; n=164, 84 | -1.0 (1.01) | -0.9 (1.03)
  Day 11; n=163, 84: number analyzed (Participants) | 163 | 84
  Day 11; n=163, 84 | -1.0 (1.05) | -0.9 (1.05)
  Day15; n=165, 84: number analyzed (Participants) | 165 | 84
  Day15; n=165, 84 | -0.9 (1.00) | -1.0 (1.03)
  Day 22; n=164, 84: number analyzed (Participants) | 164 | 84
  Day 22; n=164, 84 | -1.0 (0.99) | -1.0 (1.03)
  Day 29; n=163, 84: number analyzed (Participants) | 163 | 84
  Day 29; n=163, 84 | -1.0 (0.97) | -1.0 (1.02)
  Day 60; n=160, 83: number analyzed (Participants) | 160 | 83
  Day 60; n=160, 83 | -1.0 (1.03) | -1.0 (1.05)
  Day 90; n=160, 82: number analyzed (Participants) | 160 | 82
  Day 90; n=160, 82 | -1.0 (1.10) | -1.0 (0.96)
  Day 120; n=159, 81: number analyzed (Participants) | 159 | 81
  Day 120; n=159, 81 | -1.0 (1.05) | -0.9 (1.00)
  Day 150; n=161, 82: number analyzed (Participants) | 161 | 82
  Day 150; n=161, 82 | -1.0 (1.04) | -1.0 (1.04)
  Day180; n=160, 83: number analyzed (Participants) | 160 | 83
  Day180; n=160, 83 | -1.0 (1.04) | -1.0 (0.99)

19. Secondary Outcome: Number of Participants With P. Falciparum
Description: Microscopic blood slides (two thick film and one thin film slide) were prepared and examined for asexual parasite count. The number of participants with positive P. falciparum asexual parasite count post Baseline has been summarized for each treatment arm.
Time Frame: Up to Day 180
Population: mITT Population
Measure: Number; unit: Participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Participants | 4 | 3

20. Secondary Outcome: Number of Participants With Keratopathy
Description: Ophthalmic assessments were carried out at pre-qualified sites prior to randomization and at Days 29 and 90 and at withdrawal follow-up visit. Assessments were carried out at Day 180 (and up to resolution) if the Day 90 assessments showed abnormalities. The last assessment performed on the day of randomization or earlier was considered Baseline. The number of participants displaying keratopathy in each eye has been summarized for each visit. The number of participants with new keratopathy at any time post Baseline is also reported. Ophthalmic Safety Population comprised of all participants in the Safety Population who have results from any eye assessments. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Day 180
Population: Ophthalmic Safety Population
Measure: Number; unit: Participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 27 | 13
Participants
  Baseline; right eye; n=27, 13 | 0 | 0
  Baseline; left eye; n=27, 13 | 0 | 0
  Day 1; right eye; n=27, 13 | 0 | 0
  Day 1; left eye; n=27, 13 | 0 | 0
  Day 29; right eye; n=27, 13 | 0 | 0
  Day 29; left eye; n=27, 13 | 0 | 0
  Day 90; right eye; n=27, 12: number analyzed (Participants) | 27 | 12
  Day 90; right eye; n=27, 12 | 0 | 0
  Day 90; left eye; n=27, 12: number analyzed (Participants) | 27 | 12
  Day 90; left eye; n=27, 12 | 0 | 0
  Day 180; right eye; n=2, 2: number analyzed (Participants) | 2 | 2
  Day 180; right eye; n=2, 2 | 0 | 0
  Day 180; left eye; n=2, 2: number analyzed (Participants) | 2 | 2
  Day 180; left eye; n=2, 2 | 0 | 0
  Any time post Baseline; right eye; n=27, 13 | 0 | 0
  Any time post Baseline; left eye; n=27, 13 | 0 | 0

21. Secondary Outcome: Number of Participants With Change in Best Corrected Visual Acuity Test Scores
Description: Ophthalmic assessments were carried out at pre-qualified sites prior to randomization and at Days 29 and 90 and at withdrawal. Assessments were carried out at Day 180 if the Day 90 assessments showed abnormalities. The last assessment performed on the day of randomization or earlier was considered Baseline. Change from Baseline is the value at post dose visit minus the Baseline value. Best corrected visual acuity was assessed individually for each eye. Scores were recorded as a ratio. The values were used to derive a logMAR score for statistical analysis where logMAR=-1x log10 (ratio score). The number of participants with change in Best Corrected Visual Acuity Test Scores from Baseline has been presented where possible change is defined as a change from Baseline >=0.12 to <0.3 and definite change is defined as a change from Baseline >=0.3 logMAR score. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Day 180
Population: Ophthalmic Safety Population
Measure: Number; unit: Participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 27 | 13
Participants
  Maximum change; possible; right eye; n=27, 13 | 1 | 0
  Maximum change; definite; right eye; n=27, 13 | 0 | 0
  Maximum change; possible; left eye; n=27, 13 | 2 | 0
  Maximum change; definite; left eye; n=27, 13 | 1 | 1
  Day 29; possible change; right eye; n=27, 13 | 1 | 0
  Day 29; definite change; right eye; n=27, 13 | 0 | 0
  Day 29; possible change; left eye; n=27, 13 | 2 | 0
  Day 29; definite change; left eye; n=27, 13 | 0 | 0
  Day 90; possible change; right eye; n=27, 12: number analyzed (Participants) | 27 | 12
  Day 90; possible change; right eye; n=27, 12 | 0 | 0
  Day 90; definite change; right eye; n=27, 12: number analyzed (Participants) | 27 | 12
  Day 90; definite change; right eye; n=27, 12 | 0 | 0
  Day 90; possible change; left eye; n=27, 12: number analyzed (Participants) | 27 | 12
  Day 90; possible change; left eye; n=27, 12 | 2 | 0
  Day 90; definite change; left eye; n=27, 12: number analyzed (Participants) | 27 | 12
  Day 90; definite change; left eye; n=27, 12 | 1 | 0
  Day 180; possible change; right eye; n=2, 2: number analyzed (Participants) | 2 | 2
  Day 180; possible change; right eye; n=2, 2 | 0 | 0
  Day 180; definite change; right eye; n=2, 2: number analyzed (Participants) | 2 | 2
  Day 180; definite change; right eye; n=2, 2 | 0 | 0
  Day 180; possible change; left eye; n=2, 2: number analyzed (Participants) | 2 | 2
  Day 180; possible change; left eye; n=2, 2 | 0 | 0
  Day 180; definite change; left eye; n=2, 2: number analyzed (Participants) | 2 | 2
  Day 180; definite change; left eye; n=2, 2 | 0 | 1

22. Secondary Outcome: Number of Participants With Retinal Changes From Baseline
Description: Ophthalmic assessments were carried out at pre-qualified sites prior to randomization and at Days 29 and 90 and at withdrawal follow-up. Assessments were carried out at Day 180 (and up to resolution) if the Day 90 assessments showed abnormalities. The last assessment performed on the day of randomization or earlier was considered Baseline. Change from Baseline was calculated as the value at post dose visit minus the Baseline value. The number of participants with definite retinal change and questionable (ques) retinal change from Baseline has been presented. The number of participants with maximum change post-Baseline (definite when absent or questionable at Baseline) has been presented for either eye. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Day 180
Population: Ophthalmic Safety Population
Measure: Number; unit: Participants
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 27 | 13
Participants
  Day 29, Definite change, right eye; n=22, 13: number analyzed (Participants) | 22 | 13
  Day 29, Definite change, right eye; n=22, 13 | 0 | 0
  Day 29, Ques change, right eye; n=22, 13: number analyzed (Participants) | 22 | 13
  Day 29, Ques change, right eye; n=22, 13 | 2 | 0
  Day 29, Definite change, left eye; n=22, 13: number analyzed (Participants) | 22 | 13
  Day 29, Definite change, left eye; n=22, 13 | 0 | 0
  Day 29, Ques change, left eye; n=22, 13: number analyzed (Participants) | 22 | 13
  Day 29, Ques change, left eye; n=22, 13 | 1 | 0
  Day 90, Definite change, right eye; n=24, 11: number analyzed (Participants) | 24 | 11
  Day 90, Definite change, right eye; n=24, 11 | 0 | 0
  Day 90, Ques change, right eye; n=24, 11: number analyzed (Participants) | 24 | 11
  Day 90, Ques change, right eye; n=24, 11 | 2 | 1
  Day 90, Definite change, left eye; n=24, 11: number analyzed (Participants) | 24 | 11
  Day 90, Definite change, left eye; n=24, 11 | 0 | 0
  Day 90, Ques change, left eye; n=24, 11: number analyzed (Participants) | 24 | 11
  Day 90, Ques change, left eye; n=24, 11 | 0 | 0
  Day 180, Definite change, right eye; n=3, 2: number analyzed (Participants) | 3 | 2
  Day 180, Definite change, right eye; n=3, 2 | 0 | 0
  Day 180, Ques change, right eye; n=3, 2: number analyzed (Participants) | 3 | 2
  Day 180, Ques change, right eye; n=3, 2 | 0 | 0
  Day 180, Definite change, left eye; n=3, 2: number analyzed (Participants) | 3 | 2
  Day 180, Definite change, left eye; n=3, 2 | 0 | 0
  Day 180, Ques change, left eye; n=3, 2: number analyzed (Participants) | 3 | 2
  Day 180, Ques change, left eye; n=3, 2 | 0 | 0
  Maximum change post-Baseline; either eye; n=27, 13 | 0 | 0

23. Secondary Outcome: Change From Baseline in Percent Methemoglobin
Description: Methemoglbin is an oxidized and inactive form of hemoglobin. Methemoglobin assessment was made with the aid of a non-invasive signal extraction pulse CO-Oximeter handheld machine. The change from Baseline in percent methemoglobin by treatment, time and sex has been summarized. The latest pre-treatment assessment where treatment is their first dose of study medication (CQ/PQ/TQ/Placebo) was considered as Baseline value. Change from Baseline is the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Day 120
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | TQ+CQ | PQ+CQ
Number analyzed (Participants) | 166 | 85
Percent change
  Day 2, Male, n=114, 53: number analyzed (Participants) | 114 | 53
  Day 2, Male, n=114, 53 | 0.02 (0.754) | 0.02 (0.406)
  Day 2, Female, n=52, 32: number analyzed (Participants) | 52 | 32
  Day 2, Female, n=52, 32 | -0.16 (1.168) | -0.06 (0.181)
  Day 3, Male, n=114, 53: number analyzed (Participants) | 114 | 53
  Day 3, Male, n=114, 53 | 0.18 (0.762) | 0.03 (0.373)
  Day 3, Female, n=52, 32: number analyzed (Participants) | 52 | 32
  Day 3, Female, n=52, 32 | 0.08 (1.264) | 0.17 (0.663)
  Day 5, Male, n=113, 53: number analyzed (Participants) | 113 | 53
  Day 5, Male, n=113, 53 | 0.77 (1.226) | 0.89 (1.207)
  Day 5, Female, n=52, 32: number analyzed (Participants) | 52 | 32
  Day 5, Female, n=52, 32 | 0.63 (1.354) | 1.32 (1.400)
  Day 8, Male, n=112, 52: number analyzed (Participants) | 112 | 52
  Day 8, Male, n=112, 52 | 1.22 (1.505) | 2.63 (2.881)
  Day 8, Female, n=52, 32: number analyzed (Participants) | 52 | 32
  Day 8, Female, n=52, 32 | 1.00 (1.755) | 2.81 (2.530)
  Day 11, Male, n=112, 52: number analyzed (Participants) | 112 | 52
  Day 11, Male, n=112, 52 | 1.16 (1.446) | 3.30 (3.116)
  Day 11, Female, n=51, 32: number analyzed (Participants) | 51 | 32
  Day 11, Female, n=51, 32 | 1.04 (1.656) | 3.44 (2.651)
  Day 15, Male, n=113, 52: number analyzed (Participants) | 113 | 52
  Day 15, Male, n=113, 52 | 1.01 (1.226) | 3.26 (2.920)
  Day 15, Female, n=52, 32: number analyzed (Participants) | 52 | 32
  Day 15, Female, n=52, 32 | 0.81 (1.474) | 3.61 (2.324)
  Day 22, Male, n=112, 52: number analyzed (Participants) | 112 | 52
  Day 22, Male, n=112, 52 | 0.61 (1.008) | 1.58 (1.692)
  Day 22, Female, n=52, 32: number analyzed (Participants) | 52 | 32
  Day 22, Female, n=52, 32 | 0.32 (1.364) | 2.30 (1.900)
  Day 29, Male, n=111, 52: number analyzed (Participants) | 111 | 52
  Day 29, Male, n=111, 52 | 0.24 (0.714) | 0.46 (0.795)
  Day 29, Female, n=52, 32: number analyzed (Participants) | 52 | 32
  Day 29, Female, n=52, 32 | -0.02 (1.239) | 0.84 (0.842)
  Day 60, Male, n=107, 51: number analyzed (Participants) | 107 | 51
  Day 60, Male, n=107, 51 | 0.05 (0.583) | 0.20 (1.220)
  Day 60, Female, n=52, 32: number analyzed (Participants) | 52 | 32
  Day 60, Female, n=52, 32 | -0.09 (1.202) | 0.14 (0.496)
  Day 120, Male, n=109, 50: number analyzed (Participants) | 109 | 50
  Day 120, Male, n=109, 50 | 0.06 (0.389) | -0.01 (0.328)
  Day 120, Female, n=50, 31: number analyzed (Participants) | 50 | 31
  Day 120, Female, n=50, 31 | 0.14 (1.676) | 0.04 (0.422)

24. Secondary Outcome: Cost Associated With Relapse Episode of P Vivax Malaria
Description: Health outcomes were evaluated based on the total costs spent on treatment, transport, medication and tests. The cost was summarized according to the place at which the participant went to for care (drug shop, trial clinic, other clinic, hospital emergency center, other). The costs associated with a relapse episode of P. vivax malaria has been presented. Participants may be represented in more than one category, so the total number of participants may be less than the number quoted. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Day 180
Population: Safety Population. Only those participants who experienced a relapse or who had a follow-up visit for a relapse were included in the analysis.
Measure: Mean (Standard Deviation); unit: US Dollars (USD)
Groups:
- First Malaria Relapse: Participants from all treatment arms (CQ+TQ and PQ+TQ) with a relapse episode of malaria were included.
- First Malaria Relapse Follow-up: Participants from all treatment arms (CQ+TQ and PQ+TQ) who had a follow-up visit for relapse episode of malaria were included.
Arm/Group | First Malaria Relapse | First Malaria Relapse Follow-up
Number analyzed (Participants) | 72 | 85
US Dollars (USD)
  Brazil; enrollment clinic for care; n=19, 17: number analyzed (Participants) | 19 | 17
  Brazil; enrollment clinic for care; n=19, 17 | 8.208 (2.8369) | 8.032 (2.2403)
  Colombia; enrollment clinic for care; n=1,0: number analyzed (Participants) | 1 | 0
  Colombia; enrollment clinic for care; n=1,0 | 42.776 (0) |
  Colombia; attended another clinic; n=1,0: number analyzed (Participants) | 1 | 0
  Colombia; attended another clinic; n=1,0 | 4.194 (0) |
  Colombia; hospital emergency center; n=1,1: number analyzed (Participants) | 1 | 1
  Colombia; hospital emergency center; n=1,1 | 16.775 (0) | 16.775 (0)
  Peru; enrollment clinic for care; n=32, 33: number analyzed (Participants) | 32 | 33
  Peru; enrollment clinic for care; n=32, 33 | 9.244 (2.8235) | 8.815 (1.2803)
  Peru; attended another clinic; n=8, 30: number analyzed (Participants) | 8 | 30
  Peru; attended another clinic; n=8, 30 | 1.677 (0.9807) | 3.959 (0.8522)
  Peru; Other; n=8, 0: number analyzed (Participants) | 8 | 0
  Peru; Other; n=8, 0 | 0.818 (0.4284) |
  Thailand; enrollment clinic for care; n=0, 1: number analyzed (Participants) | 0 | 1
  Thailand; enrollment clinic for care; n=0, 1 |  | 1.534 (0)
  Vietnam; drug shop for care;n=1, 2: number analyzed (Participants) | 1 | 2
  Vietnam; drug shop for care;n=1, 2 | 0.702 (0) | 2.809 (2.6483)
  Vietnam; Other; n=1, 0: number analyzed (Participants) | 1 | 0
  Vietnam; Other; n=1, 0 | 1.873 (0) |
  Vietnam; attended another clinic; n=0, 1: number analyzed (Participants) | 0 | 1
  Vietnam; attended another clinic; n=0, 1 |  | 0.936 (0)

25. Secondary Outcome: Cost Associated With a Hemolysis Event
Description: Health outcomes were evaluated based on cost incurred due to clinically relevant hemolysis. The total cost was evaluated based on the amount spent on treatment, transport, medication and test. The costs associated with hemolysis event has been presented. The aim of this outcome measure was to determine the cost to a participant due to an event of hemolysis, regardless of treatment received in the study. It was not expected there would be major cost differences with hemoglobin decrease between the treatment arms. This was pre-specified in the statistical analysis plan.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Mean (Standard Deviation); unit: USD
Groups:
- Participants With Clinically Relevant Hemolysis: Participants from both treatment arms (TQ + CQ and PQ + CQ) with clinically relevant hemolysis were included.
Arm/Group | Participants With Clinically Relevant Hemolysis
Number analyzed (Participants) | 1
USD | 9.174 (0)

26. Secondary Outcome: Cost Incurred With Purchase of Medications Associated With Relapse Episode of P. Vivax Malaria
Description: Health outcomes were evaluated based on the cost of medications purchased. The total medication cost for paracetamol associated with relapse episode of P vivax malaria has been presented. Medications recorded as "Other" and medications without costs are excluded from the analysis. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Day 180
Population: Safety Population
Measure: Mean (Standard Deviation); unit: USD
Arm/Group | First Malaria Relapse | First Malaria Relapse Follow-up
Number analyzed (Participants) | 9 | 4
USD
  Colombia; n=2, 1: number analyzed (Participants) | 2 | 1
  Colombia; n=2, 1 | 2.516 (2.3723) | 4.194 (0)
  Peru; n=6, 2: number analyzed (Participants) | 6 | 2
  Peru; n=6, 2 | 0.491 (0.1792) | 0.327 (0.0000)
  Vietnam; n=1, 1: number analyzed (Participants) | 1 | 1
  Vietnam; n=1, 1 | 0.468 (0) | 2.341 (0)

27. Secondary Outcome: Cost Incurred With Purchase of Medications Associated With Hemolysis Event
Description: Health outcomes were evaluated based on the cost of medications purchased. The total medication cost associated with hemolysis event has been presented. Medications recorded as "Other" and medications without costs are excluded from the analysis. The aim of this outcome measure was to determine the cost to a participant due to an event of hemolysis, regardless of treatment received in the study. It was not expected there would be major cost differences with hemoglobin decrease between the treatment arms. This was pre-specified in the statistical analysis plan.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Mean (Standard Deviation); unit: USD
Arm/Group | Participants With Clinically Relevant Hemolysis
Number analyzed (Participants) | 1
USD | 0 (0)

28. Secondary Outcome: Number of Participants or Care Givers Who Had Taken Time Off From Normal Occupation Due to Relapse Episode of Malaria
Description: Health outcomes were evaluated based on total time lost by participants or care givers due to an episode of malaria. The number of participants or care givers who had taken off from their normal occupation due to relapse episode of P vivax malaria has been presented by country. Participants may be represented in more than one category, so the total number of participants may be less than the number quoted. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | First Malaria Relapse | First Malaria Relapse Follow-up
Number analyzed (Participants) | 61 | 61
Participants
  Brazil; Housework; n=2, 1: number analyzed (Participants) | 2 | 1
  Brazil; Housework; n=2, 1 | 0 | 0
  Brazil; Farming; n=1, 1: number analyzed (Participants) | 1 | 1
  Brazil; Farming; n=1, 1 | 0 | 0
  Brazil; Student; n=1, 1: number analyzed (Participants) | 1 | 1
  Brazil; Student; n=1, 1 | 0 | 0
  Brazil; Paid employment; n=7, 7: number analyzed (Participants) | 7 | 7
  Brazil; Paid employment; n=7, 7 | 0 | 0
  Brazil; Other; n=8, 7: number analyzed (Participants) | 8 | 7
  Brazil; Other; n=8, 7 | 0 | 0
  Colombia; Housework; n=1, 0: number analyzed (Participants) | 1 | 0
  Colombia; Housework; n=1, 0 | 1 |
  Colombia; Farming; n=2, 2: number analyzed (Participants) | 2 | 2
  Colombia; Farming; n=2, 2 | 0 | 0
  Colombia; Paid employment; n=1, 1: number analyzed (Participants) | 1 | 1
  Colombia; Paid employment; n=1, 1 | 1 | 1
  Peru; Housework; n=18, 18: number analyzed (Participants) | 18 | 18
  Peru; Housework; n=18, 18 | 14 | 15
  Peru, Farming; n=4, 4: number analyzed (Participants) | 4 | 4
  Peru, Farming; n=4, 4 | 4 | 4
  Peru; Student; n=3, 3: number analyzed (Participants) | 3 | 3
  Peru; Student; n=3, 3 | 2 | 2
  Peru; Paid employment; n=1, 1: number analyzed (Participants) | 1 | 1
  Peru; Paid employment; n=1, 1 | 1 | 1
  Peru; Other; n=7, 7: number analyzed (Participants) | 7 | 7
  Peru; Other; n=7, 7 | 7 | 6
  Thailand; Farming; n=1, 1: number analyzed (Participants) | 1 | 1
  Thailand; Farming; n=1, 1 | 1 | 1
  Vietnam; Farming; n=4, 4: number analyzed (Participants) | 4 | 4
  Vietnam; Farming; n=4, 4 | 3 | 1
  Vietnam; Paid employment; n=0, 3: number analyzed (Participants) | 0 | 3
  Vietnam; Paid employment; n=0, 3 |  | 2

29. Secondary Outcome: Number of Participants or Care Givers Who Had Taken Time Off From Normal Occupation Due to a Hemolysis Event
Description: Health outcomes were evaluated based on total time lost by participants or care givers due to a hemolysis event. The number of participants or care givers who took days off from work due to a hemolysis event has been presented based on the normal occupation. The aim of this outcome measure was to determine the time taken off by participants due to an event of hemolysis, regardless of treatment received in the study. It was not expected there would be major differences in time taken off by participants with hemoglobin decrease between the treatment arms. This was pre-specified in the statistical analysis plan.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Participants With Clinically Relevant Hemolysis
Number analyzed (Participants) | 1
Participants | 0

30. Secondary Outcome: Number of Participants With Action Taken to Treat Relapse Episode of P. Vivax Malaria
Description: Health outcomes were evaluated based on the actions taken by the participants to treat relapse episode of P vivax malaria. The number of participants with the type of action taken to treat relapse episode of P vivax malaria has been presented by country. Participants may be represented in more than one category, so the total number of participants may be less than the number quoted. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | First Malaria Relapse | First Malaria Relapse Follow-up
Number analyzed (Participants) | 61 | 61
Participants
  Brazil; Trial clinic; n=19, 17: number analyzed (Participants) | 19 | 17
  Brazil; Trial clinic; n=19, 17 | 19 | 17
  Brazil; Other; n=19, 17: number analyzed (Participants) | 19 | 17
  Brazil; Other; n=19, 17 | 5 | 0
  Colombia; Nothing; n=4, 3: number analyzed (Participants) | 4 | 3
  Colombia; Nothing; n=4, 3 | 2 | 2
  Colombia; Trial clinic; n=4, 3: number analyzed (Participants) | 4 | 3
  Colombia; Trial clinic; n=4, 3 | 1 | 0
  Colombia; Another clinic; n=4, 3: number analyzed (Participants) | 4 | 3
  Colombia; Another clinic; n=4, 3 | 1 | 0
  Colombia; Hospital emergency center; n=4, 3: number analyzed (Participants) | 4 | 3
  Colombia; Hospital emergency center; n=4, 3 | 1 | 1
  Peru; Trial clinic; n=33, 33: number analyzed (Participants) | 33 | 33
  Peru; Trial clinic; n=33, 33 | 32 | 33
  Peru; Another clinic; n=33, 33: number analyzed (Participants) | 33 | 33
  Peru; Another clinic; n=33, 33 | 8 | 33
  Peru; Other; n=33, 33: number analyzed (Participants) | 33 | 33
  Peru; Other; n=33, 33 | 9 | 0
  Thailand; Nothing; n=1, 1: number analyzed (Participants) | 1 | 1
  Thailand; Nothing; n=1, 1 | 1 | 0
  Thailand; Trial Clinic; n=1, 1: number analyzed (Participants) | 1 | 1
  Thailand; Trial Clinic; n=1, 1 | 0 | 1
  Vietnam; Nothing; n=4, 7: number analyzed (Participants) | 4 | 7
  Vietnam; Nothing; n=4, 7 | 1 | 5
  Vietnam; Drug Shop; n=4, 7: number analyzed (Participants) | 4 | 7
  Vietnam; Drug Shop; n=4, 7 | 2 | 2
  Vietnam; Other; n=4, 7: number analyzed (Participants) | 4 | 7
  Vietnam; Other; n=4, 7 | 1 | 0
  Vietnam; Another clinic; n=4, 7: number analyzed (Participants) | 4 | 7
  Vietnam; Another clinic; n=4, 7 | 0 | 1

31. Secondary Outcome: Number of Participants With Action Taken to Treat a Hemolysis Event
Description: Health outcomes were evaluated based on the actions taken by the participants to treat hemolysis events. The number of participants in Brazil who attended the trial clinic to treat a hemolysis event has been presented. The aim of this outcome measure was to determine the action taken by a participant due to an event of hemolysis, regardless of treatment received in the study. It was not expected there would be major differences in action taken by the participants with hemoglobin decrease between the treatment arms. This was pre-specified in the statistical analysis plan.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Participants With Clinically Relevant Hemolysis
Number analyzed (Participants) | 1
Participants | 1

32. Secondary Outcome: Oral Clearance (CL/F) of TQ
Description: Apparent population oral clearance of TQ
Time Frame: Day 2, Day 3, Day 8, Day 15, Day 29, Day 60 and Day 180
Population: Safety Population
Measure: Median (90% Confidence Interval); unit: Liters per hour
Groups:
- Participants in TQ Only Arms: TQ only arms
Arm/Group | Participants in TQ Only Arms
Number analyzed (Participants) | 166
Liters per hour | 2.96 [2.87 to 3.05]

33. Secondary Outcome: Volume of Distribution (Vc/F) of TQ
Description: Apparent population central volume of distribution of TQ
Time Frame: Day 2, Day 3, Day 8, Day 15, Day 29, Day 60 and Day 180
Population: Safety Population
Measure: Median (90% Confidence Interval); unit: Liters
Arm/Group | Participants in TQ Only Arms
Number analyzed (Participants) | 166
Liters | 915 [879 to 956]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study treatment until the follow up contact (Up to Day 180)
Description: Safety Population comprised of all randomized participants who received at least one dose of study medication.
Arm/Group | TQ+CQ | PQ+CQ
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/85
Serious Adverse Events (participants affected / at risk) | 6/166 | 1/85
Other Adverse Events (participants affected / at risk) | 97/166 | 50/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TQ+CQ (N=166) | PQ+CQ (N=85)
Haemoglobin decreased (Investigations) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TQ+CQ (N=166) | PQ+CQ (N=85)
Dizziness (Nervous system disorders) | 29 (35) | 16 (22)
Headache (Nervous system disorders) | 27 (34) | 16 (22)
Nausea (Gastrointestinal disorders) | 21 (23) | 7 (12)
Vomiting (Gastrointestinal disorders) | 15 (15) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 10 (13) | 1 (1)
Nasopharyngitis (Infections and infestations) | 14 (15) | 5 (5)
Urinary tract infection (Infections and infestations) | 9 (11) | 9 (10)
Pharyngitis (Infections and infestations) | 5 (5) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 21 (23) | 19 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (16) | 11 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 3 (4)
Pyrexia (General disorders) | 6 (7) | 6 (7)
Asthenia (General disorders) | 5 (5) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.